CLINICAL TRIAL: NCT00869947
Title: Effects of Wearing a Powered Ankle-Foot Prosthesis on Amputee Walking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: Massachusetts Institute of Technology (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: A6749-M
Record Dates: First submitted 2009-03-24; First posted 2009-03-26 (Estimated); Results first posted 2014-02-25 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-01

CONDITIONS: Traumatic Amputation of Lower Extremity
Keywords: Unilateral below the knee amputation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prosthesis (Experimental): Powered ankle-foot prosthesis and passive-elastic prosthesis
  Interventions: Device: Powered ankle-foot prosthesis
- Non-amputee (Experimental): Non-amputee
  Interventions: Other: No device

INTERVENTIONS:
Device: Powered ankle-foot prosthesis — The powered ankle-foot prosthesis is comprised of a series-elastic actuator (SEA) and an elastic leaf spring. This technology has been previously developed for robotic and human rehabilitation applications. The SEA allows for precise force control of the ankle joint, thus mimicking the spring-like behavior of the human ankle, as well as providing adequate energy for forward progression of the body. From the early stance period to the mid-stance period of walking, the SEA will be controlled so that the ankle joint behaves like a spring. During the late stance period, the SEA will be employed to power the forward movement of the body. The elastic leaf spring will provide shock absorption during foot strike, energy storage during early stance, and energy return during late stance.
  Arms: Prosthesis
Other: No device
  Arms: Non-amputee

SUMMARY:
Amputees wearing a conventional prosthesis require 20-30% more metabolic energy to walk at the same speeds as non-amputees and this discrepancy is more apparent at faster walking speeds. Amputees choose to walk at speeds 30-40% slower than non-amputees. Preferred walking speed is likely influenced by elevated metabolic energy, but the underlying reason for slower preferred walking speeds is not fully understood. Unilateral amputees exhibit highly asymmetrical gait patterns that likely require more metabolic energy and impair functional mobility, increasing the risk of degenerative joint disease, osteo-arthritis and lower back pain. Improvements in prosthetic devices could enhance mobility in amputees, thus positively effecting rehabilitation and ambulation in veterans. A prosthesis that allows amputees to reduce metabolic energy would be especially useful for rehabilitation in older, ill individuals with reduced exercise capacities and could literally restore walking ability in people that are currently non-ambulatory.

Hypotheses. Amputees wearing the Massachusetts Institute of Technology (MIT) Powered Ankle-Foot (PAF) prosthesis will have a lower metabolic cost, faster preferred walking speed, and improved gait symmetry during walking than amputees wearing a conventional prosthesis and will have nearly the same metabolic cost, preferred walking speed, and gait symmetry during walking as age, gender, height, and weight matched non-amputees.

ELIGIBILITY:
Inclusion Criteria:

* 20 healthy adult volunteers, 10 unilateral trans-tibial amputees and 10 matched non-amputees, will be recruited and screened
* Amputees must be at least 1 year post-amputation, high-functioning (at least a K3 level of ambulation), and whose cause of amputation is either traumatic or vascular. Medicare defines a K3 level amputee as an ambulator who has the ability or potential for prosthetic ambulation with variable cadence, who has the ability to traverse most environmental barriers and who may have vocational, therapeutic, or exercise activity that demands prosthetic utilization beyond simple locomotion

Exclusion Criteria:

* None

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2009-03; Primary Completion 2011-06 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alena Grabowski, PhD BA, Principal Investigator — VA Eastern Colorado Health Care System, Denver, CO
Locations (1):
- VA Medical Center, Providence, Providence, Rhode Island, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Prosthesis: Subjects with transtibial amputation using a powered and passive ankle-foot prosthesis
- Non-amputees: Non-amputees
Period: Overall Study
Arm/Group | Prosthesis | Non-amputees
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Prosthesis: Subjects with transtibial amputation using a passive ankle-foot prosthesis
- Non-amputee: Non-amputees
- Total: Total of all reporting groups
Arm/Group | Prosthesis | Non-amputee | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years]
  18 - 65 years | 46 (8) | 49 (9) | 47.5 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 8 | 8 | 16
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Metabolic Cost of Transport
Description: We measured and compared gross rates of oxygen consumption and carbon dioxide production using a portable metabolic analysis system (Cosmed K4b2, IT) while participants walked at five constance velocities (0.75, 1.00, 1.25, 1.50 and 1.75 m/s) on a level treadmill (SoleFitness F85). We calculated average steady-state metabolic power in Watts (W) from 4-6 min of each trial using a standard equation. Then, we divided the metabolic power by each participant's weight and velocity to calculate the metabolic cost of transport (J/Nm).
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: J/Nm
Arm/Group | Participants With an Amputation Using a Passive Prosthesis | Participants With an Amputation Using a Powered Prosthesis | Non-amputees
Number analyzed (Participants) | 7 | 7 | 7
J/Nm
  0.75 m/s | 4.76 (0.30) | 4.57 (0.66) | 4.68 (0.65)
  1.00 m/s | 4.11 (0.37) | 3.77 (0.31) | 3.71 (0.42)
  1.25 m/s | 3.95 (0.34) | 3.57 (0.41) | 3.41 (0.45)
  1.50 m/s | 4.15 (0.18) | 3.78 (0.34) | 3.60 (0.39)
  1.75 m/s | 4.59 (0.35) | 4.09 (0.49) | 3.69 (0.35)

2. Secondary Outcome: Preferred Walking Velocity
Description: We determined preferred walking velocity by incrementally increasing and decreasing treadmill velocity until each participant ascertained the velocity that they felt most comfortable.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Participants With an Amputation Using a Passive Prosthesis | Participants With an Amputation Using a Powered Prosthesis | Non-amputees
Number analyzed (Participants) | 7 | 7 | 7
m/s | 1.16 (0.17) | 1.42 (0.15) | 1.41 (0.25)

3. Secondary Outcome: Trailing Leg Step-to-step Transition Work
Description: We calculated step-to-step transition work, the work done by each individual leg on the center of mass during transitions, using the individual limbs method described by Donelan et al. 2002. Trailing leg step-to-step transition work quantifies the amount of push-off work done by the trailing leg when both feet are on the ground during walking. Work (J) is normalized to each subject's mass (kg).
Time Frame: 1 year
Measure: Mean (Standard Error); unit: J/kg
Arm/Group | Participants With an Amputation Using a Passive Prosthesis | Participants With an Amputation Using a Powered Prosthesis | Non-Amputees
Number analyzed (Participants) | 7 | 7 | 7
J/kg
  0.75 m/s | 0.114 (0.011) | 0.155 (0.016) | 0.165 (0.012)
  1.00 m/s | 0.125 (0.008) | 0.194 (0.013) | 0.179 (0.007)
  1.25 m/s | 0.123 (0.006) | 0.199 (0.013) | 0.199 (0.010)
  1.50 m/s | 0.131 (0.006) | 0.239 (0.017) | 0.240 (0.014)
  1.75 m/s | 0.148 (0.014) | 0.217 (0.016) | 0.259 (0.012)

ADVERSE EVENTS:
Arm/Group | Prosthesis | Non-amputees
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes